CLINICAL TRIAL: NCT07070388
Title: Robotic -Assisted Rehabilitation for Multiple Sclerosis: An Adaptive Approach for Individualized Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Holmes (Other)
Responsible Party: Sponsor-Investigator, Michael Holmes, Associate Professor, Brock University
Organization: Brock University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Brock University
Record Dates: First submitted 2025-06-27; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis
Keywords: Rehabilitation; Upper Limb; Robot; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indirect training group (Experimental): trained their self-reported less affected upper limb
  Interventions: Device: end-effector robotic training
- Direct training group (Experimental): trained their self-reported most affected limb
  Interventions: Device: end-effector robotic training

INTERVENTIONS:
Device: end-effector robotic training — For the robotic training sessions, a haptic wrist robot known as the Wristbot was used (ReWing, Genova, Italy). The training protocol consisted of an eccentric contraction-based exercise. Participants trained 3x per week for 4 consecutive weeks for approximately 25-mins per session.

SUMMARY:
Therefore, the purpose of this study was to evaluate four-weeks of an upper limb robotic intervention for persons with Multiple Sclerosis. Participants completed a resistive and adaptive robotic training intervention whereby participants trained three times weekly for four consecutive weeks.

DETAILED DESCRIPTION:
Nine individuals with Multiple Sclerosis participated and were placed into two groups based that either trained their self-reported less affected limb (indirect training group; N=4) or trained their self-reported more affected limb (direct training group; N=5).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS
* No other neurological diagnosis
* No injury to the upper limb (i.e., broken bones)

Exclusion Criteria:

- Relapse in the past 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
maximum grip force | Baseline (Week 0) and immediately post intervention (Week 4)
  Participants were asked to complete one trial of a maximum grip test (Baseline Evaluation Instruments). Held with a straight arm, 45° abduction by the side and hand/wrist neutral, participants were asked to squeeze the handle as hard as possible for 3 seconds and grip force (Newton) was recorded.
Maximum isometric wrist force | Baseline (Week 0) and immediately post intervention (Week 4)
  the participant's arm was fully extended and rested on the table, and participants were instructed to exert force at the wrist joint (F/E, RD/UD) as hard as they could against the stationary load cell that rested on the metacarpophalangeal joints (Model: BG 500, Mark-10 Corporation, New York, USA). Two maximal exertions were completed and the largest value was recorded.

SECONDARY OUTCOMES:
Wrist tracking task | Baseline (Week 0) and immediately post intervention (Week 4)
  Participants were positioned in the same position as the training. By moving the end-effector with their wrist, participants tracked a moving icon around a Lissajous-curve. Participants were instructed to follow the icon as closely as possible. The target icon moved at a velocity of 20 °/s and 5 total laps were completed. Tracking and figural error were calculated as measures of performance.
wrist range of motion | Baseline (Week 0) and immediately post intervention (Week 4)
  - Participants grasped the end-effector as target icons appeared on the monitor in front of them, participants were then asked to match the icon to the best of their abilities. When the user was at their maximal end-point range, the data was stored and recorded by the robotic device. This assessment consisted of two repetitions in each direction F/E, RD/UD.
Wolf Motor Function Test | Baseline (Week 0) and immediately post intervention (Week 4)
  functional clinical assessment of the upper limb

CONTACTS AND LOCATIONS:
Locations (1):
- Brock University, St. Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data can be made available upon request from Open-Source Journals.
Supporting Information: Study Protocol, SAP
Time Frame: June 2025 - June 2028

REFERENCES:
- [Background] Mannella, K., Albanese, G. A., Ditor, D., Zenzeri, J. & Holmes, M. W. R. Preliminary Evaluation of an Adaptive Robotic Training Program of the Wrist for Persons with Multiple Sclerosis. Appl. Sci. 11, 9239 (2021).